CLINICAL TRIAL: NCT06281899
Title: Effect of the Low PROtein Diet on Top of DAPAgliflozin and RAASi on the Progression of Chronic Kidney Disease in Patients With Type 2 Diabetes Mellitus
Brief Title: Effect of Low Protein Diet on Top of Dapagliflozin on Chronic Kidney Disease in Patients With Type 2 Diabetes Mellitus
Acronym: PRODAPA-CKD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Anemia Working Group Romania (Other)
Collaborators: Sf Ioan Emergency Clinical Hospital, Nephrology and Dialysis Department, Bucharest, Romania (Unknown); Dr Carol Davila Teaching Hospital of Nephrology, Nephrology Department, Bucharest, Romania (Unknown); Carol Davila University of Medicine and Pharmacy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01/2022
Record Dates: First submitted 2024-02-11; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Chronic Kidney Diseases; Type 2 Diabetes Mellitus
Keywords: chronic kidney disease; low protein diet; nutrition therapy
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2 | interventions — dapagliflozin; Diet, Protein-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Patients will receive a plant-based low protein diet (0.6 g proteins/kg ideal body weight per day) associated with Dapagliflozin 10 mg per day
  Interventions: Drug: Dapagliflozin 10 mg Tab; Behavioral: Low protein diet
- Control (Active Comparator): Patients will receive Dapagliflozin 10 mg per day
  Interventions: Drug: Dapagliflozin 10 mg Tab

INTERVENTIONS:
Drug: Dapagliflozin 10 mg Tab — Dapagliflozin 10 mg once daily
Behavioral: Low protein diet — Plant based low protein diet (0.6 g/kg IBW)
  Arms: Intervention

SUMMARY:
This is a prospective multicenter randomized controlled trial with a total duration of 36 months aiming to evaluate the effectiveness and the safety of low protein diet on top of sodium-glucose cotransporter 2 inhibitors (SGLT2i) and renin-angiotensin-aldosterone inhibitors (RAASi) in reducing the progression of chronic kidney disease in patients with type 2 Diabetes Mellitus

DETAILED DESCRIPTION:
The KDIGO Diabetes in CKD Guideline (2020) recommends the use of SGLT2i (level 1A) and suggests (level 2C) the prescription of plant protein-based low-protein diet in patients with chronic kidney disease (CKD) and diabetes mellitus (DM). Both interventions have shown synergistic nephroprotective effects, slowing the progression of chronic kidney disease by reducing glomerular hyperfiltration and proteinuria, thus resulting the hypothesis that by combining these two interventions it could be possible to achieve a superior control over the progression of diabetic kidney disease.

The nutritional intervention will consist in a mild protein restriction (0.6 g/kg dry ideal body weight) and a total recommended energy intake of 30-35 kcal/kg of ideal dry body weight per day in all patients. The protein intake will be checked through the food diary and calculated based on urea from 24 hours urine collection.

The efficacy and safety parameters will be evaluated during follow-up visits at month 1,2,3,6,12 and 18.

ELIGIBILITY:
Inclusion Criteria:

* age>18 years old
* confirmed chronic kidney disease (with eGFR between 60 and 20 ml/min/1.73 m2 and/or proteinuria >500 mg/g urinary creatinine) and confirmed type 2 Diabetes Mellitus
* stable kidney function for at least 12 weeks before enrollment (defined as decrease in eGFR < 5 ml/min/1.73 m2/year according to KDIGO 2012 guideline)
* treatment with ACE/ARBs and/or MRAs for at least 3 months
* no previous treatment with SGLT2i
* good nutritional status
* declared and anticipated good compliance with the prescribed diet
* signed informed consent

Exclusion Criteria:

* eGFR < 25 ml/min/1.73 m2
* poorly controlled arterial blood pressure (mean BP≥145/85 mm Hg)
* class IV NYHA heart failure, recent MACE (less than 6 months)
* relevant comorbid conditions (active infections (HBV, HCV, HIV), active neoplasia, digestive diseases with malabsorption, active autoimmune diseases/ immunosuppressive therapy)
* ADPKD
* kidney transplantation with functional graft
* malnutrition: BMI<18 kg/me, eight loss >10% during the last 6 months, serum albumin <3 g/dL
* feeding inability (anorexia, nausea)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Time to the First Occurrence of Any of the Components of the Composite: ≥30% Sustained Decline in eGFR or Reaching ESRD or CV Death or Renal Death | 12 months after randomization
  End Stage Renal Disease (ESRD) is defined as:
  * Sustained eGFR <15 mL/min/1.73m2 or,
  * Chronic dialysis treatment or,
  * Receiving a kidney transplant

SECONDARY OUTCOMES:
Rate of decline in the estimated Glomerular Filtration Rate | month 3, 9 and12 after randomization
  Difference between eGFR at any timepoint and the initial eGFR
Variation of albuminuria | month 3, 9 and12 after randomization
  Difference between albuminuria at at any timepoint and the initial albuminuria (expressed as albumin to creatinine ratio)
Variation of HbA1C | month 3, 9 and12 after randomization
  Difference between HbA1C at at any timepoint and the initial HbA1C
Variation of serum cholesterol levels | month 3, 9 and12 after randomization
  Difference between serum cholesterol at at any timepoint and the initial serum cholesterol
Variation of serum bicarbonate levels | month 3, 9 and12 after randomization
  Difference between serum bicarbonate at at any timepoint and the initial serum bicarbonate
Variation of serum potassium levels | month 3, 9 and12 after randomization
  Difference between serum potassium at at any timepoint and the initial serum potassium
Variation of serum sodium levels | month 3, 9 and12 after randomization
  Difference between serum sodium at at any timepoint and the initial serum sodium
Variation of hemoglobin levels | month 3, 9 and12 after randomization
  Difference between hemoglobin at at any timepoint and the initial serum hemoglobin
Variation of hematocrit levels | month 3, 9 and12 after randomization
  Difference between hematocrit at at any timepoint and the initial hematocrit
All cause hospitalizations | 12 months after randomization
  Percentage of patients who experienced hospitalizations of all cause
Variation in body weight | month 3, 9 and12 after randomization
  Difference between body weight at at any timepoint and the body weight
Variation in BMI | month 3, 9 and12 after randomization
  Difference between BMI at at any timepoint and the initial BMI
Variation in handgrip strength | month 3, 9 and12 after randomization
  Difference between handgrip strength at at any timepoint and the initial handgrip strength
Variation in serum albumin levels | month 3, 9 and12 after randomization
  Difference between serum albumin at at any timepoint and the initial serum albumin
Variation in CRP levels | month 3, 9 and12 after randomization
  Difference between CRP at at any timepoint and the initial CRP
Changes in the quality of life | month 3, 9 and12 after randomization
  Evaluated by SF-36 questionaire

OTHER OUTCOMES:
Compliance to the protein intake | month 1, 3, 9 and12 after randomization
  Achieved protein intake will be estimated based on urinary urea excretion, using Mitch-Maroni's formula
Compliance to the energy intake | month 1, 3, 9 and12 after randomization
  Achieved energy intake will be estimated using the 3-day food diary to calculate the daily energy intake
Compliance to carbohydrate intake | month 1, 3, 9 and12 after randomization
  Achieved energy intake will be estimated by the 3-day food diary to calculate thecarbohydrates intake

CONTACTS AND LOCATIONS:
Overall Officials: Liliana Garneata, Professor, Principal Investigator — Carol Davila University of Medicine and Pharmacy Bucharest, Romania
Locations (1):
- Carol Davila University of Medicine and Pharmacy Bucharest, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No